CLINICAL TRIAL: NCT05410626
Title: Efficacy and Safety of Generic Methylphenidate Prolong-released Comparison With Original in Child With Attention-deficit-hyperactive Disorders
Brief Title: The Study of Efficacy and Safety of Generic Methylphenidate Prolong-released Comparison With Original
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: COA.MU-DT/PY-IRB 2021/033.3003; STY.COA004/2564 (Other: Srithanya hospital)
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Adhd
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- original (Experimental): This study use 18 and 36 mg of original prolong-release methylphenidate. Dosing of Medication is equivalent to immediate-release. Medication administration is once daily in the morning.
  Interventions: Drug: prolong-release methylphenidate
- generic (Active Comparator): This study use 18 and 36 mg of generic prolong-release methylphenidate. Dosing of Medication is equivalent to immediate-release. Medication administration is once daily in the morning.
  Interventions: Drug: prolong-release methylphenidate

INTERVENTIONS:
Drug: prolong-release methylphenidate — This randomization, cross-over design study will enroll subjects who receive a stable dose of immediate-release methylphenidate (IR-MPH) for at least 4 weeks. Eligible subjects will be switching from IR-MPH to the first brand prolong-release methylphenidate (PR-MPH) for 4 weeks and switching to another brand for 4 weeks. The study consists of 3 parts: screening, study period, and post-treatment follow-up. The duration of this study will be 8 weeks with 2 visits during the study period. The primary outcome is the efficacy of treatment will be evaluated by SNAP-IV.
  Other Names: Osmotic-controlled release oral delivery system(OROS) methylphenidate, Osmotic-controlled release methylphenidate

SUMMARY:
This study is a cross-over trial, design to determine the efficacy and safety of generic and original prolong-release methylphenidate (PR-MPH) in children with ADHD who had received immediate-release methylphenidate treatment

DETAILED DESCRIPTION:
This 4 weeks cross-over study will recruit 78 children, aged 6 to 12 years, with ADHD. They will be randomized to receive generic or original PR-MPH for 4 weeks and then switch to another brand for 4 weeks. Swanson, Nolan and Pelham parent rating scale is used to measure the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 to 12 years
* Diagnosis of ADHD according to DSM-5 of ICD-10
* Patient who receiving a stable dose of IR-MPH for at least 4 weeks before screening
* Patient who has a stable clinical symptoms.
* Patients or their legal representatives provide informed consent prior to enrollment

Exclusion Criteria:

* Patients who present of a serious obstructive gastrointestinal disease
* Patients cannot swallow the whole tablet
* Patients with depression, schizophrenia, bipolar disorder, and 1-month substance use prior to study
* Patients who present of an unstable co-morbidity: anxiety, seizure, conduct disorder and oppositional defiant disorder
* Patients or patients' family have a history of poor compliance
* Patients who receiving monoamine oxidase inhibitors antidepressant or stop taking not more than 14 days
* Patients who receiving PR-MPH except stop taking more than 7 days
* Patients' parent has a family problem and currently treatment with family therapy or adjust medication

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in parent Swansan, Nolan and Pelham version IV (SNAP-IV) parent rating score | baseline, 4 and 8 week
  SNAP-IV,26 items score, included 18-items that reflect ADHD symptoms and 8-items that reflect oppositional defiant disorder symptoms

SECONDARY OUTCOMES:
The change from baseline in Clinical Global Impression-Severity (CGI-S) scale | baseline, 4 and 8 week
  CGI-S scale is measured the severity of symptoms by physician, rated from 1 (normal) to 7 (among the most severely ill patients)
The difference in discontinuation rate between two groups of treatment | 4 and 8 week
  Discontinuation rate is a proportion of patients who discontinue medication from any reason
The difference in adverse events rate between two groups of treatment | baseline, 4 and 8 week
  adverse events rate is a proportion of patients who have the adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chanatthida Muangkum, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No